CLINICAL TRIAL: NCT03735576
Title: Cognitive Behavioural Therapy for the Treatment of Late Life Depression - a Multicentre, Randomized, Observer- Blinded, Controlled Trial (CBTlate)
Brief Title: Cognitive Behavioural Therapy for the Treatment of Late Life Depression
Acronym: CBTlate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Frank Jessen, Prof. Dr., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01KG1716
Record Dates: First submitted 2018-10-24; First posted 2018-11-08 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Late-life Depression; Major Depressive Disorder; Major Depressive Episode; Major Depressive Disorder, Recurrent
Keywords: Late-life depression; Psychotherapy; Major depression; Randomized controlled trial; Treatment
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — Psychotherapy; Magnetic Resonance Spectroscopy; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Randomized, multi-center, single blind (observer-blinded), active-controlled, parallel group trial (therapeutic confirmatory) in 248 patients with late-life depression of both genders at 7 trial sites in Germany. The intervention includes 8 weeks of manual-based, individual, 15-session, twice weekly, outpatient treatment for patients with late life depression in each arm of the trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLD-adapted cognitive behavioural therapy (CBT) (Experimental): manualized 15-session individually-delivered cognitive behavioural therapy (CBT) specific for late life depression (LLD)
  Interventions: Behavioral: Psychotherapy; Diagnostic Test: Questionnaires; Other: Magnetic Resonance Imaging; Other: Blood analysis
- supportive unspecific intervention (SUI) (Active Comparator): manualized 15-session individually-delivered supportive unspecific intervention (SUI)
  Interventions: Behavioral: Psychotherapy; Diagnostic Test: Questionnaires; Other: Magnetic Resonance Imaging; Other: Blood analysis

INTERVENTIONS:
Behavioral: Psychotherapy — 15-session individually-delivered CBT specific for LLD in comparison with a supportive unspecific intervention (SUI) of the same quantity
Diagnostic Test: Questionnaires — There will be a total of four assessments (see primary & secondary endpoints). The first visit of the study will be a screening and baseline (T0) visit. After the baseline assessment, the subjects will be randomized to either of the two treatment arms. Within one week, the first of the successive bi-weekly 50-minute individual face-to-face treatment sessions will be performed by a study therapist. After 7 therapy sessions, the primary and secondary outcomes will be obtained in week 5 (T1) by the blinded rater. This will be followed by the treatment sessions 8 to 15 which will be carried out by the therapist. End-of-treatment primary and secondary outcomes will be obtained in week 10 (T2). The final follow-up assessment (T3) will be performed 6 months after randomization by the blinded rater.
Other: Magnetic Resonance Imaging — Underlying mechanisms are examined using neuroimaging. MRI data are acquired at four scanning sites and will be performed at baseline, end-of-treatment and follow-up to obtain a high-resolution structural T1-weighted image, a T2-weighted FLAIR image, a resting state fMRI, and diffusion tensor imaging (DTI) of the subjects' brain.
Other: Blood analysis — Blood sampling will be acquired in order to investigate the underlying mechanisms in LLD and the specific effects of psychotherapy. Blood samples are acquired at five sites at baseline (T0), T1, T2 and T3 for genetic and epigenetic analyses, measurement of Amyloid-β, Neurofilament light chain (NFL), Peripheral Blood Mononuclear Cells (PBMCs), Metabolomics, Proteomics and miRNA analyses.

SUMMARY:
This study addresses the unmet medical problem of insufficient treatment of late life depression (LLD). Compared with depression in early adulthood, treatment options of LLD are limited. This trial is the first confirmatory multicentre study to test the efficacy of an LLD-adapted cognitive behavioural therapy (CBT) program. It will test the hypothesis, that LLD-specific cognitive behavioural therapy (CBT) is superior to unspecific supportive intervention (SUI) with regard to reducing symptoms of depression over the course of 6 months. Secondary goals are to test the efficacy of LLD-CBT in comparison with SUI on patient reported outcome in major depressive disorders (PRO-MDD), anxiety, cognition, quality of life, overall health status, sleep and global clinical impression.

ELIGIBILITY:
Inclusion Criteria:

* out-patient status
* male or female, age ≥ 60 years
* ability to provide informed consent and written informed consent signed
* DSM-5 diagnosis of a Major Depressive Disorder/MDD (depressive episode at least moderate to severe)
* score of at least 10 on the Geriatric Depression Scale (GDS)
* score of at least 10 on the Quick Inventory of Depressive Symptomatology - Clinician Rating (QIDS-C)
* score of at least 25 in the Mini-Mental-Status-Test (MMST)
* no or stable (≥ 6 weeks) antidepressive pharmacological treatment at baseline (medication will be kept stable at least throughout the 8 weeks of treatment).
* sufficient German language skills

Exclusion Criteria:

* Bipolar depression
* Schizophrenia or other psychotic disorders
* Substance abuse or dependency
* Dementia
* Acute suicidality
* Anxiety disorder as stand-alone diagnosis (e.g. generalized anxiety disorder, panic disorder, social phobia)
* Obsessive-compulsive disorder (OCD) as stand-alone diagnosis
* Participation in any another clinical trial parallel to this trial
* Additional psychological/psychotherapeutic treatment throughout the 8-week treatment period
* Regular use with scheduled daily dosing of benzodiazepines (not PRN) during 8-week treatment
* Severe or instable medical condition, which clearly impacts on depression or on the ability to participate in the trial
* Brain disease with severe functional impairment that impacts the ability to participate in the trial (e.g. aphasia, Parkinson's disease)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Change of Geriatric Depression Scale (GDS) Score | 10 weeks
  The primary end point is the change in depression severity from baseline to week 10 measured by the 30-item Geriatric Depression Scale (GDS). It is a self-rating scale including 30 Items in a yes/no format and a total score range from 0 to 30. Higher values represent worse outcome.

SECONDARY OUTCOMES:
Change of Geriatric Depression Scale (GDS) Score | 5 weeks
  A secondary outcome measure is the change in depression severity from baseline to week 5 measured by the 30-item Geriatric Depression Scale (GDS). It is a self-rating scale including 30 Items in a yes/no format and a total score range from 0 to 30. Higher values represent worse outcome.
Change of Geriatric Depression Scale (GDS) Score | 6 months
  A secondary outcome measure is the change in depression severity from baseline to month 6 measured by the 30-item Geriatric Depression Scale (GDS). It is a self-rating scale including 30 Items in a yes/no format and a total score range from 0 to 30. Higher values represent worse outcome.
Change of Quick Inventory of Depressive Symptomatology Score - Clinician Rating (QIDS-C) | 5 weeks
  A secondary outcome measure is the change in depression severity from baseline to week 5 measured by the 16-item Quick Inventory of Depressive Symptomatology Score - Clinician Rating (QIDS-C). It is a clinician-rated scale including 16 Items and a total score range from 0 to 27. Higher values represent worse outcome.
Change of Quick Inventory of Depressive Symptomatology Score - Clinician Rating (QIDS-C) | 10 weeks
  A secondary outcome measure is the change in depression severity from baseline to week 10 measured by the 16-item Quick Inventory of Depressive Symptomatology Score - Clinician Rating (QIDS-C). It is a clinician-rated scale including 16 Items and a total score range from 0 to 27. Higher values represent worse outcome.
Change of Quick Inventory of Depressive Symptomatology Score - Clinician Rating (QIDS-C) | 6 months
  A secondary outcome measure is the change in depression severity from baseline to month 6 measured by the 16-item Quick Inventory of Depressive Symptomatology Score - Clinician Rating (QIDS-C). It is a clinician-rated scale including 16 Items and a total score range from 0 to 27. Higher values represent worse outcome.
Change of Patient Reported Outcome for Major Depressive Disorder (PRO-MDD) Score | 10 weeks
  A secondary outcome measure is the change in depression severity from baseline to week 10 measured by the 35-item Patient Reported Outcome for Major Depressive Disorder (PRO-MDD) Score. It is a self-rating scale including 35 Items on an11-point numeric rating scale. Higher values represent worse outcome.
Change of Patient Reported Outcome for Major Depressive Disorder (PRO-MDD) Score | 6 months
  A secondary outcome measure is the change in depression severity from baseline to month 6 measured by the 35-item Patient Reported Outcome for Major Depressive Disorder (PRO-MDD) Score. It is a self-rating scale including 35 Items on an11-point numeric rating scale. Higher values represent worse outcome.
Longitudinal Interval Follow-up Evaluation (LIFE) | 6 months
  A secondary outcome measure is the longitudinal evaluation of depressive symptoms by the Longitudinal Interval Follow-up Evaluation Interview (LIFE) at month 6.
Change of Insomnia Severity Index (ISI) Score | 10 weeks
  A secondary outcome measure is the change in insomnia severity from baseline to week 10 measured by the 7-item Insomnia Severity Index (ISI). It is a self-rating scale including 7 Items rated on a scale from 0 to 4 from less to more severe. The total score ranges from 0 to 28. Higher values represent worse outcome.
Change of Insomnia Severity Index (ISI) Score | 6 months
  A secondary outcome measure is the change in insomnia severity from baseline to month 6 measured by the 7-item Insomnia Severity Index (ISI). It is a self-rating scale including 7 Items rated on a scale from 0 to 4 from less to more severe. The total score ranges from 0 to 28. Higher values represent worse outcome.
Change of Epworth Sleepiness Scale (ESS) Score | 10 weeks
  A secondary outcome measure is the change in sleepiness from baseline to week 10 measured by the 8-item Epworth Sleepiness Scale (ESS). It is a self-rating scale including 8 Items rated on a 4-point Likert scale. The total score ranges from 0 to 24. Higher values represent worse outcome.
Change of Epworth Sleepiness Scale (ESS) Score | 6 months
  A secondary outcome measure is the change in sleepiness from baseline to month 6 measured by the 8-item Epworth Sleepiness Scale (ESS). It is a self-rating scale including 8 Items rated on a 4-point Likert scale. The total score ranges from 0 to 24. Higher values represent worse outcome.
Change of REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ)Score | 10 weeks
  A secondary outcome measure is the change in REM sleep behavior from baseline to week 10 measured by the 10-item REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ). It is a self-rating scale including 10 Items in a yes/no format. The total score ranges from 0 to 13. Higher values represent worse outcome.
Change of REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ)Score | 6 months
  A secondary outcome measure is the change in REM sleep behavior from baseline to month 6 measured by the 10-item REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ). It is a self-rating scale including 10 Items in a yes/no format. The total score ranges from 0 to 13. Higher values represent worse outcome.
Change of Geriatric Anxiety Inventory (GAI) Score | 10 weeks
  A secondary outcome measure is the change in anxiety symptoms from baseline to week 10 measured by the 20-item Geriatric Anxiety Inventory (GAI). It is a self-rating scale including 20 Items in a agree/disagree format and a total score range from 0 to 20. The cut-off score of 9 classifies the presence of clinically significant anxiety. Higher values represent worse outcome.
Change of Geriatric Anxiety Inventory (GAI) Score | 6 months
  A secondary outcome measure is the change in anxiety symptoms from baseline to month 6 measured by the 20-item Geriatric Anxiety Inventory (GAI). It is a self-rating scale including 20 Items in a agree/disagree format and a total score range from 0 to 20. The cut-off score of 9 classifies the presence of clinically significant anxiety. Higher values represent worse outcome.
Change in Quality of Life (WHOQOL) | 10 weeks
  A secondary outcome measure is the change in quality of life from baseline to week 10 measured by the 24-item WHOQOL-OLD and 26-item WHOQOL-BREF.
Change in Quality of Life (WHOQOL) | 6 months
  A secondary outcome measure is the change in quality of life from baseline to month 6 measured by the 24-item WHOQOL-OLD and 26-item WHOQOL-BREF.
Change in Short Form Health Survey (SF-36) | 10 weeks
  A secondary outcome measure is the change in overall health status from baseline to week 10 measured by the 36-item Short Form Health Survey (SF-36).
Change in Short Form Health Survey (SF-36) | 6 months
  A secondary outcome measure is the change in overall health status from baseline to month 6 measured by the 36-item Short Form Health Survey (SF-36).
Change in Subjective Cognitive Functioning | 6 months
  A secondary outcome measure is the change in subjective cognitive functioning from baseline to month 6 measured by the semi-structured Subjective Cognitive Decline interview.
Change in cognitive function (CERAD-Plus) | 6 months
  A secondary outcome measure is the change in cognitive function from baseline to month 6 measured by the Consortium to Establish a Registry for Alzheimer's Disease (CERAD-Plus) neuropsychological test battery.
Change in executive function (NAB maze test) | 6 months
  A secondary outcome measure is the change in executive function from baseline to month 6 measured by the Neuropsychological Assessment Battery (NAB) maze subtest.
Childhood Trauma Questionnaire (CTQ) | baseline
  Assessment of the severity of five categories of childhood trauma(emotional/physical/sexual abuse and emotional/physical neglect) at baseline
Big Five-Inventory 10 Item Short Version (BFI-10) | baseline
  10-item scale measuring the personality traits Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness to assess the influence of personality traits on treatment outcome at baseline. The items are rated on a five-step scale from 1 "disagree strongly" to 5 "agree strongly". The scale consists of 2 BFI items for each Big Five Dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jessen, Prof.Dr., Principal Investigator — University of Cologne
Locations (7):
- Germany (7):
  - Charité Berlin, Berlin
  - University of Bonn, Bonn
  - University of Cologne, Cologne
  - University of Freiburg, Freiburg im Breisgau
  - University of Leipzig, Leipzig
  - ZI Mannheim, Mannheim
  - University of Tuebingen, Tübingen

REFERENCES:
- [Derived] Bewernick B, Buschmann J, Heser K, Kleineidam L, Domschke K, Elsaesser M, Zehender N, Luppa M, Hellmich M, Peters O, Froelich L, Riedel-Heller S, Schramm E, Hautzinger M, Jessen F, Dafsari FS, Wagner M. The effect of cognition and age on the efficacy of psychotherapy in late-life depression. J Affect Disord. 2025 Dec 15;391:119881. doi: 10.1016/j.jad.2025.119881. Epub 2025 Jul 14. PMID 40669702
- [Derived] Dafsari FS, Bewernick B, Bohringer S, Domschke K, Elsaesser M, Lobner M, Luppa M, Schmitt S, Wingenfeld K, Wolf E, Zehender N, Hellmich M, Muller W, Wagner M, Peters O, Frolich L, Riedel-Heller S, Schramm E, Hautzinger M, Jessen F. Perceived Physical Health and Cognitive Behavioral Therapy vs Supportive Psychotherapy Outcomes in Adults With Late-Life Depression: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245841. doi: 10.1001/jamanetworkopen.2024.5841. PMID 38619842
- [Derived] Dafsari FS, Bewernick B, Biewer M, Christ H, Domschke K, Froelich L, Hellmich M, Luppa M, Peters O, Ramirez A, Riedel-Heller S, Schramm E, Vry MS, Wagner M, Hautzinger M, Jessen F. Cognitive behavioural therapy for the treatment of late life depression: study protocol of a multicentre, randomized, observer-blinded, controlled trial (CBTlate). BMC Psychiatry. 2019 Dec 27;19(1):423. doi: 10.1186/s12888-019-2412-0. PMID 31881995